CLINICAL TRIAL: NCT01682148
Title: A Phase III Prospective, Multi-center, Randomised, Evaluator-blinded Study to Compare Neuromuscular Junction (NMJ) Targeted Technique for Dysport Injections in Upper Limb Spasticity Post Stroke or Traumatic Brain Injury to the Technique Used in Current Clinical Practice
Brief Title: Comparing Lower-concentration Dysport Treatment Targeted to the Neuromuscular Junction With Current Clinical Practice
Acronym: NMJ
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to slow recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-99-52120-162; 2011-005375-16 (EudraCT Number)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Arm Spasticity
Keywords: Dysport; arm spasticity; Modified Ashworth Scale; neuromuscular junction; Botulinum toxin; upper limb spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMJ Targeted (Experimental): NMJ targeted technique and low-concentration dilution (Dysport 100 U/mL). The same number and sites of injections/deposits per muscle were given as per prestudy. With a Dysport dilution of 300 U/mL the volume to be injected varied between 0.1 mL and 0.7 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
  Interventions: Biological: Botulinum toxin type A
- Current Clinical Practice (Active Comparator): Current clinical practice technique and high-concentration dilution (Dysport 300 U/mL).
  A single injection per muscle was given in the midline of the band of NMJ zones. With a Dysport dilution of 100 U/mL the volume to be injected varied between 0.4 mL and 2.0 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The aim of the study was to compare Dysport treatment results (as assessed by Modified Ashworth Scale (MAS) in the elbow joint 4 weeks post treatment) following two treatment techniques: the current clinical practice injection technique using high-concentration dilution (300 U/mL Dysport) versus the neuromuscular junction (NMJ)-targeted injection technique using low-concentration dilution (100 U/mL Dysport). The hypothesis was that one high-volume, low-concentration injection located centrally in the area/band of the NMJ zones would be as effective as the technique used in current medical practice.

DETAILED DESCRIPTION:
This was a randomised, evaluator-blinded, comparative, parallel group, multicentre study, conducted in four countries (Denmark, Finland, Norway and Sweden). For each subject, the primary efficacy assessments using MAS were performed by the same blinded evaluator, and every effort was made at each site to ensure that the MAS evaluator was the same person throughout the study. Dysport doses were to follow clinical practice for subjects suffering from upper limb spasticity position pattern type 1, 3 or 4 post stroke or traumatic brain injury.

The hypothesis for this study was that one low-concentration botulinum neurotoxin type A (BoNT-A) injection per muscle, centrally located in the area/band of the NMJ zones, would spread to and block the surrounding NMJ zones and be as effective as the technique used today in clinical practice. The possibility to reduce the number of injection points would decrease the risk of injection discomfort, pain and injection site bleeding for the patient. A simplified injection technique with one injection per muscle and in a defined location would also benefit physicians.

At Baseline (Visit 1), subjects were randomised to one of two treatment groups:

* Group 1: Current clinical practice technique and high-concentration dilution: Dysport 300 U/mL.
* Group 2: NMJ targeted technique and low-concentration dilution: Dysport 100 U/mL.

Each subject visited the clinic on at least three occasions:

* Baseline (Visit 1): Screening, randomisation and Dysport treatment.
* Week 4 (Visit 2): Treatment follow-up, 4 weeks after Dysport treatment.
* Week 12 (Visit 3): Treatment and study follow-up, 12 weeks after Dysport treatment.

For subjects not receiving any post study BoNT-A injection at Week 12 due to remaining treatment effect, an extra visit (Visit 4) for study follow-up was to take place at the next routine visit planned for a new BoNT-A injection, at the latest 24 weeks post study injection.

The duration of each subject's study period was at a minimum 12 weeks and maximum 24 weeks. The overall duration of the study was planned to be approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* Subjects male or female, aged 18 years or older.
* Upper limb spasticity post stroke or traumatic brain injury.
* Spasticity position pattern type 1, 3 or 4.
* Elbow flexor muscles spasticity MAS 2 to 3.
* At least 2 consecutive previous treatment cycles of BoNT-A for current diagnosis.
* The latest treatment cycle demonstrating good treatment efficacy where the Dysport dose administered was considered to be adequate according to Investigator judgement.
* Need of the same treatment modality in muscle (m.) brachialis, m. biceps brachii, m. brachioradialis, m. flexor carpi ulnaris, m. flexor carpi radialis as the previous treatment cycle.
* Last BoNT-A treatment 12-24 weeks ago.

Exclusion Criteria:

* Poor response to BoNT-A treatment, according to Investigator.
* Need of Dysport doses >800 U in the upper limb.
* Concomitant treatment with BoNT-A for other indications than spasticity.
* Any elbow flexor contracture prohibiting MAS evaluation and/or elbow flexion improvement of at least 1 step on the MAS.
* Cutaneous or joint inflammation in the affected upper limb.
* Was likely to start other spasticity treatment during the study.
* Was likely to start physiotherapy treatment during the study.
* Other ongoing neurological disorder (e.g., myasthenia gravis).
* History of dysphagia or aspiration.
* Use of agents interfering with neuromuscular transmission (e.g., aminoglycosides).
* Treated with an investigational medicinal product within 30 days before start of the study.
* Known sensitivity to BoNT-A or any components of Dysport.
* Was at risk of pregnancy or was lactating. Females of childbearing potential must have provided a negative pregnancy test (urinary human chorionic gonadotropin (U-hCG)) at Visit 1 and must have been using adequate contraception. Non-childbearing potential was defined as post-menopause for at least one year, surgical sterilisation or hysterectomy at least three months before the start of the study.
* Had a history of, or known current, problems with alcohol or drug abuse.
* Had a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* Had abnormal Baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might have jeopardised the subject's safety or decreased the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (23):
- Denmark (7):
  - Aalborg Sygehus Nord, Aalborg
  - Glostrup Hospital, Glostrup Municipality
  - Regionshospitalet Hammel, Hammel
  - Bispebjerg Hospital, København NV
  - Roskilde Hospital, Roskilde
  - Vejle Hospital, Vejle
  - Regionshopsitalet Viborg, Viborg
- Finland (2):
  - North Karelia Central Hospital, Joensuu
  - Central Hospital of Central Finland, Jyväskylä
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Sykehuset Telemark HF, Skien
- Sweden (12):
  - Mälarsjukhuset MSE, Eskilstuna
  - Sahlgrenska University Hospital, Gothenburg
  - Hallands Sjukhus, Neurology Clinic, Halmstad
  - Sundsvall-Härnösand, Rehabilitation Medicine, Härnösand
  - Nyköpings Lasarett,, Nyköping
  - Örnsköldsviks Sjukhus, Neurology Clinic, Örnsköldsvik
  - Östersunds Rehabilitation Center, Östersund
  - Neurorehab Sävar, Sävar
  - Neurology Clinic Stockholm, Stockholm
  - Danderyds Hospital,, Stockholm
  - Rehabilitation Center Gotland, Visby
  - Ystad Lasarett, Ystad

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Rekand T, Biering-Sorensen B, He J, Vilholm OJ, Christensen PB, Ulfarsson T, Belusa R, Strom T, Myrenfors P, Maisonobe P, Dalager T. Botulinum toxin treatment of spasticity targeted to muscle endplates: an international, randomised, evaluator-blinded study comparing two different botulinum toxin injection strategies for the treatment of upper limb spasticity. BMJ Open. 2019 May 5;9(5):e024340. doi: 10.1136/bmjopen-2018-024340. PMID 31061021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2012, subjects were recruited across 20 sites in four countries: Denmark (5 sites), Finland (2 sites), Norway (2 sites) and Sweden (11 sites). Due to slow recruitment, the study was terminated early.
Pre-assignment Details: 272 subjects were planned to be randomised (136 subjects in each group). In total, 100 subjects were enrolled and 88 (44 subjects in each group) were randomised and received study medication; 12 subjects were screening failures.
Groups:
- NMJ Targeted: Neuromuscular junction (NMJ) targeted technique and low-concentration dilution (Dysport 100 U/mL): A single injection per muscle was given in the midline of the band of NMJ zones. With a Dysport dilution of 100 U/mL the volume to be injected varied between 0.4 mL and 2.0 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
- Current Clinical Practice: Current clinical practice technique and high-concentration dilution (Dysport 300 U/mL): The same number and sites of injections/deposits per muscle were given as per prestudy. With a Dysport dilution of 300 U/mL the volume to be injected varied between 0.1 mL and 0.7 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
Period: Overall Study
Arm/Group | NMJ Targeted | Current Clinical Practice
Started | 44 | 44
Completed | 40 | 41
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population was defined as all treated subjects having at least one Baseline assessment of the primary efficacy parameter. The ITT population was analysed using subjects as randomised.
Groups:
- NMJ Targeted: NMJ targeted technique and low-concentration dilution (Dysport 100 U/mL): A single injection per muscle was given in the midline of the band of NMJ zones. With a Dysport dilution of 100 U/mL the volume to be injected varied between 0.4 mL and 2.0 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
- Total: Total of all reporting groups
Arm/Group | NMJ Targeted | Current Clinical Practice | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Customized [Mean (Standard Deviation); unit: years] | 57.1 (11.4) | 60.3 (14.4) | 58.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 30 | 28 | 58
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 17 | 17 | 34
  Norway | 2 | 3 | 5
  Finland | 5 | 5 | 10
  Denmark | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Elbow Flexors Muscle Tone as Measured by the Modified Ashworth Scale (MAS) at Week 4
Description: A clinically relevant change was one level decrease on the MAS scale. Subjects meeting the defined decrease at Week 4 were considered as responders in the primary efficacy analysis.
Time Frame: Baseline to Week 4
Population: The primary analysis was based on both the ITT and Per Protocol (PP) populations. The ITT population was all treated subjects having at least one Baseline assessment of the primary efficacy parameter. The PP population was all subjects in the ITT population for whom no major protocol violations or deviations occurred until Week 4 (Visit 2).
Measure: Number; unit: responders
Groups:
- NMJ Targeted (ITT Population); NMJ Targeted (PP Population): NMJ targeted technique and low-concentration dilution (Dysport 100 U/mL): A single injection per muscle was given in the midline of the band of NMJ zones. With a Dysport dilution of 100 U/mL the volume to be injected varied between 0.4 mL and 2.0 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
- Current Clinical Practice (ITT Population); Current Clinical Practice (PP Population): Current clinical practice technique and high-concentration dilution (Dysport 300 U/mL): The same number and sites of injections/deposits per muscle were given as per prestudy. With a Dysport dilution of 300 U/mL the volume to be injected varied between 0.1 mL and 0.7 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment.
Arm/Group | NMJ Targeted (ITT Population) | Current Clinical Practice (ITT Population) | NMJ Targeted (PP Population) | Current Clinical Practice (PP Population)
Number analyzed (Participants) | 44 | 44 | 25 | 29
responders | 25 | 32 | 17 | 20
Statistical Analysis 1: Comparison: NMJ Targeted (ITT Population) vs Current Clinical Practice (ITT Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — Based on a responder rate (π) of 63% in the reference group, a clinically relevant delta (Δ) of 17%, α=2.5% (one sided) and power=80%, the sample size estimate yielded 122 valid subjects per group. Including a 10% addition for premature withdrawals, 136 subjects per group were necessary to be randomised in the study (i.e., a total of 272 subjects); p = 0.0986, Generalised linear model — Based on a generalised linear model including factors for treatment; Treatment difference = -0.1673, 95% CI 2-sided [-0.3630 to 0.0284] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 2: Comparison: NMJ Targeted (ITT Population) vs Current Clinical Practice (ITT Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — Based on a π of 63% in the reference group, a clinically relevant Δ of 17%, α=2.5% (one sided) and power=80%, the sample size estimate yielded 122 valid subjects per group. Including a 10% addition for premature withdrawals, 136 subjects per group were necessary to be randomised in the study (i.e., a total of 272 subjects); p = 0.5682, Generalised linear model — Based on a generalised linear model including factors for spasticity pattern; Treatment difference = -0.1673, 95% CI 2-sided [-0.3630 to 0.0284] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 3: Comparison: NMJ Targeted (ITT Population) vs Current Clinical Practice (ITT Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.8543, Generalised linear model — Based on a generalised linear model including factors for country; Treatment difference = -0.1673, 5% CI 2-sided [-0.3630 to 0.0284] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 4: Comparison: NMJ Targeted (ITT Population) vs Current Clinical Practice (ITT Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.9167, Generalised linear model — Based on a generalised linear model including factors for MAS at Baseline; Treatment difference = -0.1673, 95% CI 2-sided [-0.3630 to 0.0284] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 5: Comparison: NMJ Targeted (PP Population) vs Current Clinical Practice (PP Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.6052, Generalised linear model — Based on a generalised linear model including factors for treatment; Treatment difference = 0.0707, 95% CI 2-sided [-0.1948 to 0.3362] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 6: Comparison: NMJ Targeted (PP Population) vs Current Clinical Practice (PP Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.5369, Generalised linear model — Based on a generalised linear model including factors for spasticity pattern; Treatment difference = 0.0707, 95% CI 2-sided [-0.1948 to 0.3362] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 7: Comparison: NMJ Targeted (PP Population) vs Current Clinical Practice (PP Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.7732, Generalised linear model — Based on a generalised linear model including factors for country; Treatment difference = 0.0707, 95% CI 2-sided [-0.1948 to 0.3362] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)
Statistical Analysis 8: Comparison: NMJ Targeted (PP Population) vs Current Clinical Practice (PP Population); A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.1758, Generalised linear model — Based on a generalised linear model including factors for MAS at Baseline; Treatment difference = 0.0707, 95% CI 2-sided [-0.1948 to 0.3362] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)

2. Secondary Outcome: Change From Baseline for Elbow Flexors Muscle Tone as Measured by the Modified Ashworth Scale (MAS) at Week 4 and Week 12
Description: Increased muscle tone in elbow flexors was assessed using the MAS. Scale ranges from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension).
Time Frame: Baseline to Week 12
Population: ITT population: all treated subjects having at least one Baseline assessment of the primary efficacy parameter. Only subjects with non-missing values were included in this analysis.
  CCP=Current Clinical Practice; N'=number of subjects with data at each time point for each treatment group; NMJ=neuromuscular junction.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 40 | 43
units on a scale
  Baseline to Week 4 | -0.5 [-2 to 1] | -1.0 [-3 to 1]
  Baseline to Week 12: number analyzed (Participants) | 39 | 39
  Baseline to Week 12 | 0.0 [-2 to 1] | 0.0 [-2 to 1]

3. Secondary Outcome: Change From Baseline for Elbow Flexors Muscle Tone as Measured by the MAS at Week 12
Description: A clinically relevant change was one level decrease on the MAS scale. Subjects meeting the defined decrease at Week 12 were considered as responders.
Time Frame: Baseline to Week 12
Population: ITT population: all treated subjects having at least one Baseline assessment of the primary efficacy parameter. Only subjects with non-missing values were included in the analysis.
Measure: Number; unit: responders
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 39 | 39
responders | 13 | 19
Statistical Analysis 1: Comparison: NMJ Targeted vs Current Clinical Practice; A responder was defined as a subject with at least one level decrease on the MAS scale; Test type: Superiority or Other; p = 0.2400, Generalised linear model — Based on a generalised linear model including factors for treatment, spasticity pattern, country and MAS baseline score; Treatment difference = -0.1324, 95% CI 2-sided [-0.3531 to 0.0884] — Difference of the two clinical success rates (NMJ Targeted minus Current Clinical Practice)

4. Secondary Outcome: Change From Baseline of Spasticity Related Pain Measured by Visual Analogue Scale (VAS), Assessed by the Subject
Description: Pain assessment using the VAS. The VAS was a 10 cm straight horizontal line scoring scale. Score range on VAS was from 0 to 10 where 0 indicated no pain and 10 indicated worst pain imaginable.
Time Frame: Baseline, Week 4 and Week 12
Population: ITT population: all treated subjects having at least one Baseline assessment of the primary efficacy parameter.
  CCP=Current Clinical Practice; N'=number of subjects with data at each time point for each treatment group; NMJ=neuromuscular junction.
Measure: Mean (Standard Deviation); unit: Change in VAS from Baseline
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 44 | 44
Change in VAS from Baseline
  Week 4: number analyzed (Participants) | 40 | 43
  Week 4 | -5.80 (23.07) | -4.35 (12.29)
  Week 12: number analyzed (Participants) | 39 | 39
  Week 12 | -0.03 (26.02) | 0.03 (20.67)
Statistical Analysis 1: Comparison: NMJ Targeted vs Current Clinical Practice; Mean change in VAS from Baseline to Week 4; Test type: Superiority or Other; p = 0.9448, ANOVA; Analysis of variance (ANOVA) included factors for treatment, spasticity pattern and country, and Baseline VAS as a covariate
Statistical Analysis 2: Comparison: NMJ Targeted vs Current Clinical Practice; Mean change in VAS from Baseline to Week 12; Test type: Superiority or Other; p = 0.5458, ANOVA; ANOVA included factors for treatment, spasticity pattern and country, and Baseline VAS as a covariate

5. Secondary Outcome: Injection Site Pain Measured by VAS at Day 1.
Description: Pain assessment using the VAS. The VAS was a 100 mm straight horizontal line scoring scale. Score range on VAS was from 0 to 100 where 0 indicated no pain and 100 indicated worst pain imaginable.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 36 | 37
mm | 25.67 (25.37) | 30.68 (27.33)
Statistical Analysis 1: Comparison: NMJ Targeted vs Current Clinical Practice; Test type: Superiority or Other; p = 0.4006, ANOVA; ANOVA included factors for treatment, spasticity pattern and country

6. Secondary Outcome: Achievement of the Primary Goal Measured by Goal Attainment Scale (GAS)
Description: At Baseline, an agreed primary goal related to elbow flexion in one of the following categories was determined: active function, impairment, involuntary movement, mobility, pain passive function or other. Each goal was usually rated -1, unless the subject was as bad as he/she could be in that particular goal area, in which case the Baseline score was -2. The evaluator rated the outcome score at Week 4 or Week 12, depending on the time point defined at the baseline visit (Visit 1), using the GAS five-point scale (-2, -1, 0, +1 and +2).
Time Frame: Up to Week 12
Population: ITT population: all treated subjects having at least one Baseline assessment of the primary efficacy parameter. Only subjects with non-missing values were included in the analysis. Only overall GAS score data are summarised below.
Measure: Count of Participants; unit: Participants
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 33 | 41
Participants
  Overall GAS score of -2 | 3 | 1
  Overall GAS score of -1 | 9 | 15
  Overall GAS score of 0 | 11 | 18
  Overall GAS score of +1 | 9 | 6
  Overall GAS score of +2 | 1 | 1
Statistical Analysis 1: Comparison: NMJ Targeted vs Current Clinical Practice; Test type: Superiority or Other; p = 0.5747, Mann-Whitney U-test

7. Secondary Outcome: Subject Global Evaluation of Treatment Effect
Description: Comparison of treatment effect between previous (prestudy) and study treatment cycles assessed by the subject at the end of study (Week 12 up to Week 24 (Visit 3 or Visit 4)). Categorised as follows: Much worse / Worse / Same / Better / Much better.
Time Frame: Up to Week 24
Population: ITT population: all treated subjects having at least one Baseline assessment of the primary efficacy parameter. Only subjects with non-missing values were included in the analysis. If a subject had more than one evaluation entry, the last one was used.
Measure: Count of Participants; unit: Participants
Arm/Group | NMJ Targeted | Current Clinical Practice
Number analyzed (Participants) | 40 | 40
Participants
  Much Better | 3 | 2
  Better | 11 | 16
  No Change From Baseline | 18 | 20
  Worse | 7 | 2
  Much Worse | 1 | 0
Statistical Analysis 1: Comparison: NMJ Targeted vs Current Clinical Practice; Test type: Superiority or Other; p = 0.1802, Mann-Whitney U-test

8. Secondary Outcome: Investigator Preference of Injection Technique
Description: When all patients at the site had completed the study (last subject last visit) a global assessment of the injection technique was to be made by the Investigators. The following question was answered: "Based on your experience during this study, which injection technique do you prefer?"
Time Frame: Following last visit of the last subject at each site
Population: The question on preferred injection technique was answered by 3 of the 20 Investigators.
Measure: Number; unit: Investigators
Groups:
- Number of Investigators Who Responded: Investigator preference for using the NMJ Targeted versus the Current Clinical Practice technique was requested at each of the 20 sites (20 Investigators).
Arm/Group | Number of Investigators Who Responded
Number analyzed (Participants) | 3
Investigators
  NMJ Targeted | 1
  Current Clinical Practice | 2

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored from informed consent to the time when the subject's participation in the study ended (Week 12 to Week 24 (Visit 3 or Visit 4)). AEs were elicited by direct, non-leading questioning at each clinic visit or by spontaneous reports.
Description: The safety population was defined as all subjects who received at least one dose of study medication. The safety population was analysed using subjects as treated. If a subject experienced more than one event in a System Organ Class (SOC), the subject was counted only once in that SOC.
Groups:
- Current Clinical Practice: Current clinical practice technique and high-concentration dilution (Dysport 300 U/mL): The same number and sites of injections/deposits per muscle were given as per prestudy. With a Dysport dilution of 300 U/mL the volume to be injected varied between 0.1 mL and 0.7 mL per muscle. The dose and the choice of muscles involved in the elbow flexion were the same as for the last prestudy treatment .
Arm/Group | NMJ Targeted | Current Clinical Practice
Serious Adverse Events (participants affected / at risk) | 2/44 | 2/44
Other Adverse Events (participants affected / at risk) | 13/44 | 9/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NMJ Targeted (N=44) | Current Clinical Practice (N=44)
Cystitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NMJ Targeted (N=44) | Current Clinical Practice (N=44)
Headache (Nervous system disorders) | 3 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site hypersensitivity (General disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to slow recruitment, the study was terminated early. Therefore, fewer subjects than planned were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor required reasonable opportunity to review any abstract, presentation or paper before the material was submitted for publication or communicated. This also applied to any amendments that were requested by referees or journal editors. The Sponsor committed to comment on the draft documents within the time period agreed in the contractual arrangements between the Sponsor and authors or their institution. Delays were also possible if publication would adversely affect patentability.